CLINICAL TRIAL: NCT04807530
Title: Causal Role of Medial Prefrontal Neural Activity in Self-Agency in Schizophrenia
Brief Title: Medial-prefrontal Enhancement During Schizophrenia Systems Imaging
Acronym: MESSI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122897; 1R01MH122897-01 (NIH)
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Transcranial Magnetic Stimulation; Prefrontal Cortex; Self-Agency; Reality Monitoring
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: The investigators propose a longitudinal randomized controlled trial (RCT) in which 80 SZ and 80 HC are randomly assigned to either active high-frequency 10Hz nrTMS to increase activity in medial/superior prefrontal cortex (mPFC) or a control posterior parietal site. The investigators assess durability and generalizability of how active 10Hz nrTMS modulation of mPFC activity in HC and SZ causally induces neural network changes that mediate behavioral changes in self-agency to impact overall cognition, clinical and daily functioning, compared to the control parietal site and baseline.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and care providers and all clinical outcomes assessors will be blinded as to whether participants will receive the active nrTMS or control nrTMS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Medial/Superior Prefrontal TMS (Active Comparator): 10 Hz High frequency TMS applied to the mPFC
  Interventions: Device: TMS
- Posterior Parietal TMS (Placebo Comparator): 10 Hz high frequency TMS applied to the posterior parietal cortex
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — The investigators will use the NEXSTIM NAVIGATED BRAIN STIMULATION (NBS) SYSTEM to apply 10 Hz nrTMS to healthy controls (HC) and schizophrenia patients (SZ)

SUMMARY:
This randomized controlled trial in healthy controls (HC) and patients with schizophrenia (SZ) aims to examine 1) the underlying cognitive and neural cause of self-agency deficits in SZ; 2) the responsiveness to a novel navigated repetitive transcranial magnetic stimulation (nrTMS) target in the medial/superior prefrontal cortex (mPFC); and 3) how modulation of mPFC activity impacts the larger self-agency network to mediate changes in self-agency judgments. Our overall hypothesis is that increased mPFC excitability by active high-frequency nrTMS in HC and SZ will induce behavioral improvements in self-agency and neural changes in the larger self-agency network that will generalize to improvements in overall cognition, symptoms and daily functioning, and will likely lead to the development of new effective neuromodulation therapies in patients with schizophrenia.

DETAILED DESCRIPTION:
This longitudinal mechanistic randomized controlled trial in patients with schizophrenia (SZ) and matched healthy controls (HC) examines the underlying cause of self-agency deficits in SZ and their responsiveness to navigated repetitive transcranial magnetic stimulation (nrTMS) of the medial prefrontal cortex. Using a multimodal neuroimaging approach that combines structural MRI with functional magnetoencephalography imaging (MEGI) and nrTMS that is integrated with cognitive and clinical assessments, this research provides an unprecedented rigorous assessment of the neural and cognitive basis of self-agency and its modulation by nrTMS, using two distinct and validated paradigms involving speech monitoring (pitch perturbation) and reality monitoring.

Subjects will first be assessed for 1 week for diagnostic inclusion criteria and eligibility assessment. They will complete baseline assessments (i.e., cognitive, clinical and daily functioning assessments, structural MRI, and MEGI scans while they perform reality and speech monitoring tasks). After baseline assessments, 80 SZ and 80 age, gender, and education-matched HC will be randomly assigned to either active 10Hz nrTMS targeting mPFC (40HC and 40SZ) or nrTMS targeting a control posterior parietal site (40HC and 40SZ). For the parietal site, the investigators will use the same TMS protocol parameters as the active nrTMS condition. Between and within group analyses will utilize repeated measures mixed-effects models to examine durability and generalizability of behavioral, cognitive, clinical and whole-brain neural oscillatory network changes (with focus on mPFC) after neuromodulation by active nrTMS at proximal, and distal post-nrTMS time-points, compared to control nrTMS of parietal site and baseline. Whole-brain correlations will be computed between neural activity (e.g., with focus on mPFC) related to self-agency during reality and speech monitoring tasks and behavior (e.g., self-generated retrieval accuracy and corrective response magnitude), and between neural activity with cognition, clinical symptoms and daily functioning).

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Good general physical health
* English is first language
* No neurological disorder
* Meets MRI criteria
* No current alcohol or substance use disorder

Schizophrenia participants:

* Schizophrenia diagnosis of any illness duration,
* Clinical stability, defined as 12 weeks outpatient status and 4 weeks low to moderate dose of antipsychotic medication (<1000 mg. chlorpromazine equivalents), plus stable doses of all other psychotropic medications

Exclusion Criteria:

All Subjects:

* Implanted metallic parts of implanted electronic devices
* Pregnant or trying to become pregnant
* Any condition that would prevent the subject from giving voluntary informed consent
* Scalp wounds or infections
* Claustrophobia precluding MRI
* Ongoing seizures
* Neurological disorder

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-Agency Behavioral Change during Reality Monitoring after TMS vs Baseline (metrics of accuracy) | From baseline, to immediately after TMS, up to 1 week
  Change in retrieval accuracy of self-generated information during reality monitoring task from baseline to post-TMS. No scales used.
Self-Agency Behavioral Change during Speech Monitoring after TMS vs Baseline (metrics of speech perturbation units) | From baseline, to immediately after TMS, up to 1 week
  Change in speech corrective responses during altered vs. unaltered auditory feedback, measured in units of speech perturbation (cents) from baseline to post-TMS. No scales used.
MEGI Neural Activity Change related to Self-Agency during Reality Monitoring after TMS vs Baseline (metrics of neural beta activation units) | From baseline, to immediately after TMS, up to 1 week
  Whole-brain neural activity change related to self-agency by contrasting oscillatory activity during encoding and retrieval of self-generated information with encoding and retrieval of externally-derived information (with focus on mPFC and parietal cortices as our region-of-interest (ROI)), measured in beta weights neural signal change from baseline to post-TMS. No scales used.
MEGI Neural Activity Change related to Self-Agency during Speech Monitoring after TMS vs Baseline (metrics of neural beta activation units) | From baseline, to immediately after TMS, up to 1 week
  Whole-brain neural activity related to self-agency by contrasting oscillatory activity related to speech onset during altered auditory feedback with activity related to speech onset during unaltered auditory feedback (with focus on mPFC and parietal cortices for ROI analyses) measured in beta weights neural signal change from baseline to post-TMS. No scales used.

SECONDARY OUTCOMES:
Cognition Change after TMS vs Baseline (metrics units of accuracy and speed of processing) | From baseline to immediate and distal time points after TMS, up to 4 weeks
  The PENN Cognitive battery is a validated assessment of cognition in which accuracy scores and reaction times will computed after TMS compared to baseline.The PENN Cognitive battery includes 10 brief cognitive tests, and the score ranges between 0 (worst possible performance) and 1000 (best possible performance).
Clinical Symptom Change after TMS vs Baseline (metrics units of severity) | From baseline to immediate and distal time points after TMS, up to 4 weeks
  Clinical Symptom Change will be measured by the validated SAPS and SANS over the past week after TMS compared to baseline. Possible scores depending on the sub scale can range from 0(Absent) to 7 (Extreme).
Daily Functioning Change after TMS vs. Baseline (metrics of functioning) | From baseline to immediate and distal time points after TMS, up to 4 weeks
  Daily functioning will be measured with the Global Assessment of Functioning (GAF) scale over the past week, after TMS compared to baseline. Possible score range from 0 (inadequate information or in persistent danger of severely hurting self or others) to 100 (superior functioning in a wide range of activities)

CONTACTS AND LOCATIONS:
Overall Officials: Karuna Subramaniam, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will include clinical, behavioral and cognitive scores, nrTMS data, and neuroimaging data. Neuroimaging data will include MEGI and structural MRI scans. All de-identified data will also be made available through presentations at scientific conferences, symposia, and seminars, as well as through publications in scientific journals. All University of California employees are committed to an open access policy to make all publications freely available. In compliance with this policy, all publications resulting from this proposal will be submitted for archiving on PubMed Central and BioRxiv.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators aim to complete all data analyses by end of 2025-2026, when the complete, and all deidentified data will be available for sharing